CLINICAL TRIAL: NCT00738673
Title: An Open-Label, Multi-Centre, Uncontrolled, Exploratory Trial Investigating Degarelix One-Month Dosing Regimen as Second-Line Hormonal Treatment After PSA-Failure in GnRH Agonist Treated Patients With Prostate Cancer
Brief Title: Degarelix as Second-Line Hormonal Treatment After Prostate-specific Antigen (PSA)-Failure in GnRH Agonist Treated Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS27; 2008-000585-22 (EudraCT Number)
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: Hormone refractory prostate cancer; Agonist treatment failure
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental): Starting dose: 240 mg by subcutaneous (s.c.) injection in the abdomen on Day 0.
  Maintenance dose: a maximum of 11 doses of 80 mg degarelix were given 28 days apart via single s.c. injections.
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix — Starting dose of 240 mg (40 mg/mL). Maintenance doses of 80 mg (20 mg/mL).
  Other Names: FE200486

SUMMARY:
This was an open-label, multi-centre, uncontrolled, exploratory trial with a duration of 12 months in two cohorts. The trial aimed to investigate Degarelix as a second-line hormonal treatment in Prostate Cancer patients who experienced PSA-Failure following gonadotropin-releasing hormone (GnRH) agonist treatment. The two cohorts differ in Testosterone levels at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent before any trial-related activity is performed.
* Patient is 18 years or older.
* Histologically confirmed prostate cancer.
* Patient has received GnRH receptor agonist therapy for a duration of at least 12 months (the first dose of GnRH-antagonist is to be administered when the next dose of the GnRH-agonist would have been due).
* Patient has experienced rising PSA levels although receiving GnRH agonist therapy, defined as two consecutive rises of PSA at least two weeks apart in two 50% increases over the nadir, and at least one PSA value of >2.5 ng/mL within the last six months.
* Testosterone on castrate level (defined as ≤ 0.5 ng/mL) (cohort 1); Testosterone ≥0.2 ng/mL at inclusion (cohort 2)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Estimated life expectancy at least 12 months.

Exclusion Criteria:

* Previous history or presence of another malignancy, other than prostate cancer or treated squamous / basal cell carcinoma of the skin, within the last five years.
* Ongoing GnRH agonist therapy (last dose of previous GnRH agonist must have been received before Visit 1).
* Any pre-trial secondary hormonal manipulation (including antiandrogens) after PSA increase as described as above and before trial entry. Antiandrogens as part of complete androgen blockade must have been discontinued at least three months before first dose of trial medication.
* Previous or current treatment with chemotherapy (e.g. estramustine) for prostate cancer.
* Known hypersensitivity towards any component of the investigational medical product.
* History of severe uncontrolled asthma, anaphylactic reactions, or severe urticaria and/or angioedema.
* Known or suspected clinically significant liver and/or biliary disease.
* Any clinically significant laboratory abnormalities, disorders, or other condition, including alcohol or drug abuse, which may affect the patient's health or the outcome of the trial as judged by the Investigator.
* Patient has a clinically significant disorder (other than prostate cancer) including, but not limited to, renal, hematological, gastrointestinal, endocrine, cardiac, neurological, or psychiatric disease, and alcohol or drug abuse or any other condition, which may affect the patient's health or the outcome of the trial as judged by the Investigator.
* Patient has a mental incapacity or language barriers precluding adequate understanding or co-operation.
* Patient has received an investigational drug within the last 28 days preceding screening visit. Or longer if considered to possibly influencing the outcome of the current trial.
* Previous participation in any degarelix trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (15):
- Germany (15):
  - Urologische Praxis, Bautzen
  - Urologische Klinik, Berlin
  - Urologische Praxis, Berlin
  - Urologische Praxis, Borken
  - Urologische Praxis, Cologne
  - Urologische Praxis, Erkrath - Hochdal
  - Urologische Praxis, Hagenow
  - Martini Klinik, Hamburg
  - Urologische Praxis, Husum
  - Urologische Praxis, Kirchheim
  - Urologische Praxis, Lauenburg/Elbe
  - Urologische Praxis, Leipzig
  - Urologische Praxis, Markkleeberg
  - Urologische Klinik, Planegg
  - Wissenschaftskontor Nord, Rostock

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 comprised a broad spectrum of biochemically relapsed participants (on castrate level) on long term hormonal treatment in different stages of the disease (primarily advance stages), however not in need of chemotherapy. The second cohort was similar, although testosterone levels were to be above castrate level (≥0.32 ng/mL).
Groups:
- Degarelix - Cohort 1: Participants with baseline testosterone at castrate level. Starting dose: 240 mg by subcutaneous (s.c.) injection in the abdomen on Day 0. Maintenance dose: a maximum of 11 doses of 80 mg degarelix were given 28 days apart via single s.c. injections.
- Degarelix - Cohort 2: Participants with baseline testosterone above castrate level (≥0.32 ng/mL ). Starting dose: 240 mg by subcutaneous (s.c.) injection in the abdomen on Day 0. Maintenance dose: a maximum of 11 doses of 80 mg degarelix were given 28 days apart via single s.c. injections.
Period: Overall Study
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Started | 25 | 12
Intent to Treat Population | 24 | 12
Completed | 1 | 1
Not Completed | 24 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 19 | 8
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2 | Total
Number analyzed (Participants) | 24 | 12 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 72.7 (9.11) | 76.5 (4.68) | 73.9 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 12 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 24 | 12 | 36
  HIspanic or Latino | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24 | 12 | 36
  Other | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 90.5 (17.3) | 87.6 (11.0) | 89.6 (15.5)
Height [Mean (Standard Deviation); unit: meters] | 1.74 (0.06) | 1.72 (0.05) | 1.73 (0.06)
Stage of Prostate Cancer at Diagnosis [Number; unit: participants]
  Localized | 4 | 4 | 8
  Locally advanced | 11 | 1 | 12
  Metastatic | 6 | 2 | 8
  Not classifiable | 3 | 5 | 8
Stage of Prostate Cancer at Enrolment [Number; unit: participants]
  Localized | 1 | 2 | 3
  Locally advanced | 9 | 0 | 9
  Metastatic | 7 | 5 | 12
  Not classifiable | 7 | 5 | 12
Gleason Score [Number; unit: participants] — The 2005 International Society of Urological Pathologists recommendations for Gleason scoring were used to grade tumors. A primary grade is assigned to the most common tumor pattern (how the cancer cells look under a microscope), and a second grade to the next most common pattern. The two grades are added together to get a Gleason Score with a range of 2-10; 10=worst prognosis.
  participants
    2-4 | 1 | 3 | 4
    5-6 | 4 | 2 | 6
    7-10 | 19 | 7 | 26
Eastern Cooporative Oncology Group (ECOG) Performance Status [Number; unit: participants]
  Fully active | 0 | 0 | 0
  Restricted, but ambulatory | 17 | 11 | 28
  Ambulatory, unable to work | 7 | 1 | 8
  Capable of only limited selfcare | 0 | 0 | 0
  Completely disabled | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants' Response in Prostate-Specific Antigen (PSA) Level at Three Months As Compared to Baseline
Description: Response to treatment was defined as:
  * Response (stabilisation or decrease): Difference ≤ +10% of Baseline level
  * No response (increase): Difference > +10% of Baseline level
Time Frame: Day 0 (baseline), 3 months
Population: Intent to treat population. Last observation carried forward.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 24 | 12
percentage of participants
  Response | 16.67 [4.74 to 37.38] | 33.33 [9.92 to 65.11]
  No Response | 83.33 [62.62 to 95.26] | 66.67 [34.89 to 90.08]

2. Secondary Outcome: Participants' Response in Prostate-Specific Antigen (PSA) Level at One Month As Compared to Baseline
Description: Response to treatment was defined as:
  * Response (stabilisation or decrease): Difference ≤ +10% of Baseline level
  * No response (increase): Difference > +10% of Baseline level.
  Per protocol, the one month timeframe was only analyzed for cohort 2.
Time Frame: Day 0 (baseline), 1 month
Population: Full analysis set of participants with baseline and month 1 values. Per protocol, the one month timeframe was only analyzed for cohort 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 0 | 9
percentage of participants
  Response |  | 66.67 [29.93 to 92.51]
  No Response |  | 33.33 [7.49 to 70.07]

3. Secondary Outcome: Participants' Response in Prostate-Specific Antigen (PSA) Level at Two Months As Compared to Baseline
Description: Response to treatment was defined as:
  * Response (stabilisation or decrease): Difference ≤ +10% of Baseline level
  * No response (increase): Difference > +10% of Baseline level.
  Per protocol, the two month timeframe was only analyzed for cohort 2.
Time Frame: Day 0 (baseline), 2 months
Population: Full analysis set of participants with baseline and month 2 values. Per protocol, the two month timeframe was only analyzed for cohort 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 0 | 10
percentage of participants
  Response |  | 40.00 [12.16 to 73.76]
  No Response |  | 60.00 [26.24 to 87.84]

4. Secondary Outcome: Participants at Testosterone Castrate Level Throughout the Study
Description: Participants who had no post-baseline serum testosterone level above castrate level which was <=0.5 ng/mL.
Time Frame: up to month 12
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 24 | 12
participants | 24 | 11

5. Secondary Outcome: Change From Baseline in Serum Levels of Testosterone at the Last Visit
Time Frame: Day 0 (baseline), up to month 12 (last visit)
Population: Intent to treat population with a baseline and at least one scheduled post-baseline measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 24 | 9
ng/mL | -0.039 (0.175) | -0.038 (0.631)

6. Secondary Outcome: Change From Baseline in Serum Levels of Prostate-Specific Antigen (PSA) at Last Visit
Time Frame: Day 0 (baseline), up to month 12 (last visit)
Population: Intent to treat population with a baseline and at least one scheduled post-baseline measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 24 | 9
ng/mL | 18 (29) | 54 (116)

7. Secondary Outcome: Percent Change From Baseline in Serum Levels of Luteinising Hormone (LH) at the Last Visit
Description: LH is measured in IU/L
Time Frame: Day 0 (baseline), up to month 12 (last visit)
Population: Intent to treat population with a baseline and at least one scheduled post-baseline measurement.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 24 | 9
percentage of baseline | 58 (286) | 123 (277)

8. Secondary Outcome: Change From Baseline in Serum Levels of Follicle-Stimulating Hormone (FSH) at the Last Visit
Time Frame: Day 0 (baseline), up to month 12 (last visit)
Population: Intent to treat population with a baseline and at least one scheduled post-baseline measurement.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 24 | 9
IU/L | -1.64 (3.01) | -2.01 (1.72)

9. Secondary Outcome: Participants at Testosterone Level <=0.2 ng/mL Throughout the Study
Description: Participants in Cohort 2 who had no post-baseline serum testosterone level above 0.2 ng/mL.
Time Frame: up to month 12
Population: Full analysis set. Per the protocol, this analysis was only performed on Cohort 2.
Measure: Number; unit: participants
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 0 | 12
participants |  | 8

10. Secondary Outcome: Participants at Testosterone Level <=0.32 ng/mL Throughout the Study
Description: Participants in Cohort 2 who had no post-baseline serum testosterone level above 0.32 ng/mL
Time Frame: up to month 12
Population: Full analysis set. Per the protocol, this analysis was only performed on Cohort 2.
Measure: Number; unit: participants
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 0 | 12
participants |  | 9

11. Secondary Outcome: Participants With Prostate-Specific Antigen (PSA) Progression Throughout the Study
Description: Counts of participants who had PSA progression during the study. PSA progression was defined as PSA >+10% of baseline value.
Time Frame: up to month 12
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 24 | 12
participants | 21 | 11

12. Secondary Outcome: Kaplan-Meier Estimate for Overall Survival
Description: The overall survival time was defined as number of days from first treatment dose to date of death. If a patient did not die then the patient's data were censored at the date of last visit.
Time Frame: up to month 12
Population: Intent to treat population.
  Analysis was not performed since no participants died during study.
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to month 13
Arm/Group | Degarelix - Cohort 1 | Degarelix - Cohort 2
Serious Adverse Events (participants affected / at risk) | 3/25 | 1/12
Other Adverse Events (participants affected / at risk) | 18/25 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix - Cohort 1 (N=25) | Degarelix - Cohort 2 (N=12)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix - Cohort 1 (N=25) | Degarelix - Cohort 2 (N=12)
Constipation (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Injection site erythema (General disorders) | 10 | 6
Injection site swelling (General disorders) | 8 | 5
Injection site pain (General disorders) | 3 | 0
Injection site induration (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Weight increase (Investigations) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hot flush (Vascular disorders) | 2 | 0
Venous stasis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.